CLINICAL TRIAL: NCT03383809
Title: Impact of Non Digestible Carbohydrate on Production of Phenolic Acids From Strawberry Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Scottish Universities Environmental Research Centre (Other)
Responsible Party: Principal Investigator, Christine Edwards, Professor, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BB/MO27724/1-1
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Self-reported healthy adults
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Intervention Model Description: Acute human bioavailability studies with a cross-over design will be given to subjects in the form of a drink in one of three combinations
  1. Strawberry juice alone
  2. Inulin alone
  3. Mixture of strawberry juice and inulin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strawberry juice with inulin (Experimental): One dose of 300 g of strawberry with 10 g of inulin will be given to subjects in the form of juice
  Interventions: Dietary Supplement: Strawberry juice with Inulin
- Strawberry juice (Experimental): One dose of 300 g of strawberry juice will be given to subjects in the form of juice
  Interventions: Dietary Supplement: Strawberry Juice
- Inulin (Experimental): One dose of 10 g of inulin will be given to subjects in the form of a drink
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Strawberry juice with Inulin — Mixture of polyphenols and non digestible carbohydrates
  Arms: Strawberry juice with inulin
Dietary Supplement: Strawberry Juice — Source of Polyphenols
  Arms: Strawberry juice
Dietary Supplement: Inulin — Source of non digestible carbohydrate
  Arms: Inulin

SUMMARY:
This is an acute human bioavailability study in self-reported healthy participants aged 20-70 years old. We hypothesize that combination of dietary polyphenolics and non-digestible carbohydrates (NDC) will increase the production of phenolic acids by bacteria in the human colon and these will be detected in urine. Participants will attend for three arms in a randomised order: Strawberry juice (a high polyphenol food), Inulin (NDC) or Mixture of strawberry juice and inulin.

DETAILED DESCRIPTION:
Polyphenol rich plant foods have been associated with several health benefits but their bioavailability is generally low. The majority of plant polyphenols are poorly absorbed in the small intestine and enter the colon where the colonic microbiota metabolise them to release a range of phenolic acids, which are now thought to be the main bioactive components related to the reduction in disease risk. Very little is known about the impact of other constituents of the diet on the metabolism and bacterial catabolism of these polyphenols. The colonic microbiota are key agents in the release of the bioactive molecules from polyphenols but also ferment non-digestible carbohydrates (NDC) such as dietary fibre to short chain fatty acids. It is likely that there are key interactions in the colonic bacteria metabolism of fibre and phenolics. We hypothesize that combination of polyphenolics and non-digestible carbohydrates (NDC) will increase the urinary output of bioactive phenolic acids.

This study will enable a better understanding of how to deliver combinations of ingredients and nutrients to achieve maximum nutritional value and health benefits.

ELIGIBILITY:
Inclusion Criteria:

Self-reported healthy adults

Exclusion Criteria:

Antibiotic use within the last 3 months, identified gastro-intestinal diseases, on prescribed medication other than the contraceptive pill, individuals who are pregnant or breastfeeding. Individuals who have been diagnosed as anaemic, as well as those who are allergic to any food, or paracetamol.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
Phenolic acids bioavailability | 0-24 hrs
  Urine excretion of phenolic acids

SECONDARY OUTCOMES:
Urolithin bioavailability | 0-24 hrs
  Urine excretion of urolithins
Glycaemic and appetite hormones measurements by ELISA | 0-8 hrs
  Plasma glucose, insulin and appetite hormone levels
Mouth to caecum transit time | 0-8 hrs
  Breath hydrogen level measurements by Hydrogen monitor
Gastric emptying time | 0-6 hrs
  Plasma paracetamol levels by acetaminophen assay kits

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Edwards, Principal Investigator — University of Glasgow
Locations (1):
- School of Medicine, Nursing and Dentistry, College of MVLS, University of Glasgow, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- [Background] Russell W, Duthie G. Plant secondary metabolites and gut health: the case for phenolic acids. Proc Nutr Soc. 2011 Aug;70(3):389-96. doi: 10.1017/S0029665111000152. PMID 21781364
- [Background] Roowi S, Mullen W, Edwards CA, Crozier A. Yoghurt impacts on the excretion of phenolic acids derived from colonic breakdown of orange juice flavanones in humans. Mol Nutr Food Res. 2009 May;53 Suppl 1:S68-75. doi: 10.1002/mnfr.200800287. PMID 19415668
- [Background] Henning SM, Wang P, Abgaryan N, Vicinanza R, de Oliveira DM, Zhang Y, Lee RP, Carpenter CL, Aronson WJ, Heber D. Phenolic acid concentrations in plasma and urine from men consuming green or black tea and potential chemopreventive properties for colon cancer. Mol Nutr Food Res. 2013 Mar;57(3):483-93. doi: 10.1002/mnfr.201200646. Epub 2013 Jan 14. PMID 23319439
- [Background] Czank C, Cassidy A, Zhang Q, Morrison DJ, Preston T, Kroon PA, Botting NP, Kay CD. Human metabolism and elimination of the anthocyanin, cyanidin-3-glucoside: a (13)C-tracer study. Am J Clin Nutr. 2013 May;97(5):995-1003. doi: 10.3945/ajcn.112.049247. PMID 23604435
- [Background] Morrison DJ, O'Hara JP, King RF, Preston T. Quantitation of plasma 13C-galactose and 13C-glucose during exercise by liquid chromatography/isotope ratio mass spectrometry. Rapid Commun Mass Spectrom. 2011 Sep 15;25(17):2484-8. doi: 10.1002/rcm.5139. PMID 21818809